CLINICAL TRIAL: NCT02547766
Title: Interleukin-1 Receptor Antagonist for the Treatment of Heart Failure in Patients With Left Ventricular Assist Devices
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Craig Selzman, M.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 75500
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Ventricular Assist Device; Recovery of Function
MeSH Terms: conditions — Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra Arm (Experimental): All patients in this arm receive Anakinra in a pre-post design. That is, outcome markers are measured, the intervention (Anakinra) is applied, and the outcome markers are measured again at various intervals to determine effect.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra is an Interleukin-1 receptor antagonist that will be given to the patient via subcutaneous injection for a period of 14 consecutive days.
  Other Names: Kineret

SUMMARY:
Heart failure remains a major cause of morbidity and mortality. Many patients with heart failure receive support from a left ventricular assist device (LVAD) at some point in the course of their disease. Some of these LVAD patients experience a durable recovery after ventricular unloading with an LVAD, which may be associated with inhibition of inflammatory cytokines. This small pilot study aims to determine the biologic and clinical efficacy of an interleukin-1 receptor antagonist (Anakinra) at inducing myocardial recovery in patients supported with left ventricular assist devices.

DETAILED DESCRIPTION:
More than 5 million Americans have heart failure, a number that is expected to increase 25% by the year 2030. Fifty percent of individuals diagnosed with heart failure die within 5 years of diagnosis. Of those patients who currently have heart failure, 5-10% have Stage D disease, requiring specialized interventions such as chronic inotropic support, mechanical circulatory support, or transplantation. Transplantation is considered curative for heart failure, but only about 2,200 heart transplants take place each year. Due to the imbalance between donors and possible recipients, a large number of patients remain who could benefit from transplantation that will never receive a heart. Many patients receive left ventricular assist devices (LVADs) to support their failing hearts, increasing their chances of survival while they wait to undergo transplantation.

It has been shown that up to 19% of patients show durable echocardiographic recovery (as measured by left ventricular ejection fraction >40%) after ventricular unloading with an LVAD. Recovery mediated by unloading with the LVAD causes several changes at the molecular level. However, the mechanisms underlying recovery at the cellular level, also known as reverse remodeling, are only recently being studied. Thus, the window of opportunity to develop adjuvant treatments to enhance recovery is just now opening.

Interestingly, patients that experience durable echocardiographic recovery have higher circulating levels of anti-inflammatory cytokines. Inhibition of inflammatory cytokines, such as with the use of receptor antagonists for inflammation-associated cytokines like Anakinra, has also been shown to reduce adverse myocardial remodeling after ischemic events and to increase exercise activity in patients with systolic heart failure. This study proposes the exogenous administration of Anakinra to end-stage heart failure patients supported with LVADs in an effort to increase both the number of patients who experience recovery and the magnitude of recovery.

While this is a small trial aimed primarily at demonstrating biologic efficacy of Anakinra, clinical efficacy in this study is also investigated. Encouraging results in this pilot study may prompt the creation of a randomized, controlled trial designed to demonstrate efficacy from a functional clinical standpoint.

ELIGIBILITY:
Inclusion Criteria:

* To qualify for inclusion, patients must meet the following criteria: age >18 years at date of LVAD implantation who require circulatory support with an LVAD for either a bridge-to-transplant or destination therapy indication.
* They must also be judged by the implanting surgeon to have an expected survival to trial completion (approximately 6 months after implantation), without regard to the likelihood of cardiac transplantation.

Exclusion Criteria:

* Exclusion criteria include the presence of a Right Ventricular Assist Device, as biventricular support is associated with decreased survival outcomes that could negatively impact the attrition rate over the course of the study.
* Additional exclusion criteria include the inability of the patient or a trained caregiver to administer the study drug, and inability of the patient to complete the study questionnaire. - Patients with a creatinine clearance < 30 mL/min, evidence of an active infection, immunosuppression, or with an allergy to E. Coli derived products will also be excluded. -
* Last, any patient with dependence on inflammatory modulating drugs will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Birks EJ, Tansley PD, Hardy J, George RS, Bowles CT, Burke M, Banner NR, Khaghani A, Yacoub MH. Left ventricular assist device and drug therapy for the reversal of heart failure. N Engl J Med. 2006 Nov 2;355(18):1873-84. doi: 10.1056/NEJMoa053063. PMID 17079761
- [Background] Abbate A, Van Tassell BW, Biondi-Zoccai G, Kontos MC, Grizzard JD, Spillman DW, Oddi C, Roberts CS, Melchior RD, Mueller GH, Abouzaki NA, Rengel LR, Varma A, Gambill ML, Falcao RA, Voelkel NF, Dinarello CA, Vetrovec GW. Effects of interleukin-1 blockade with anakinra on adverse cardiac remodeling and heart failure after acute myocardial infarction [from the Virginia Commonwealth University-Anakinra Remodeling Trial (2) (VCU-ART2) pilot study]. Am J Cardiol. 2013 May 15;111(10):1394-400. doi: 10.1016/j.amjcard.2013.01.287. Epub 2013 Feb 27. PMID 23453459
- [Background] Abbate A, Kontos MC, Grizzard JD, Biondi-Zoccai GG, Van Tassell BW, Robati R, Roach LM, Arena RA, Roberts CS, Varma A, Gelwix CC, Salloum FN, Hastillo A, Dinarello CA, Vetrovec GW; VCU-ART Investigators. Interleukin-1 blockade with anakinra to prevent adverse cardiac remodeling after acute myocardial infarction (Virginia Commonwealth University Anakinra Remodeling Trial [VCU-ART] Pilot study). Am J Cardiol. 2010 May 15;105(10):1371-1377.e1. doi: 10.1016/j.amjcard.2009.12.059. Epub 2010 Apr 2. PMID 20451681
- [Background] Drakos SG, Wever-Pinzon O, Selzman CH, Gilbert EM, Alharethi R, Reid BB, Saidi A, Diakos NA, Stoker S, Davis ES, Movsesian M, Li DY, Stehlik J, Kfoury AG; UCAR (Utah Cardiac Recovery Program) Investigators. Magnitude and time course of changes induced by continuous-flow left ventricular assist device unloading in chronic heart failure: insights into cardiac recovery. J Am Coll Cardiol. 2013 May 14;61(19):1985-94. doi: 10.1016/j.jacc.2013.01.072. Epub 2013 Mar 14. PMID 23500219
- [Background] Drakos SG, Kfoury AG, Selzman CH, Verma DR, Nanas JN, Li DY, Stehlik J. Left ventricular assist device unloading effects on myocardial structure and function: current status of the field and call for action. Curr Opin Cardiol. 2011 May;26(3):245-55. doi: 10.1097/HCO.0b013e328345af13. PMID 21451407
- [Background] Guglin M, Miller L. Myocardial recovery with left ventricular assist devices. Curr Treat Options Cardiovasc Med. 2012 Aug;14(4):370-83. doi: 10.1007/s11936-012-0190-9. PMID 22760582
- [Derived] Healy AH, Bowen M, McKellar SH, Koliopoulou A, Drakos SG, Selzman CH. Interleukin-1 Receptor Antagonism as Adjunct Therapy for Heart Failure Patients with Left Ventricular Assist Devices. ASAIO J. 2021 Aug 1;67(8):e145-e147. doi: 10.1097/MAT.0000000000001347. PMID 33470637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra Arm
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Biologic Efficacy: Inflammation Marker - C-Reactive Protein
Description: The primary endpoint was a reduction in inflammatory markers, specifically C-reactive protein (CRP).
Time Frame: 6 months post treatment
Population: Patients
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Anakinra Arm
Number analyzed (Participants) | 10
mg/dL
  Prior to Anakinra | 2.5 [1.1 to 3.0]
  After Anakinra | 0.6 [0.4 to 1.8]
  At 6 months | 0.6 [0.5 to 1.7]

2. Secondary Outcome: Biologic Efficacy: Inflammation Marker - Neutrophil Count
Description: Secondary endpoints included the measure of additional inflammatory markers, including neutrophil count.
Time Frame: 6 months post treatment
Population: Patients
Measure: Median (Full Range); unit: 10^3 cells/µL
Arm/Group | Anakinra Arm
Number analyzed (Participants) | 10
10^3 cells/µL
  Prior to Anakinra | 6.4 [5.7 to 6.7]
  After Anakinra | 5.0 [2.8 to 5.4]
  At 6 months | 4.4 [3.6 to 5.3]

3. Secondary Outcome: Clinical Efficacy: Ejection Fraction
Description: Clinical efficacy was a secondary endpoint that was measured using ejection fraction (EF)
Time Frame: 6 months post treatment
Population: Patients
Measure: Median (Full Range); unit: percentage of blood leaving heart
Arm/Group | Anakinra Arm
Number analyzed (Participants) | 10
percentage of blood leaving heart
  Prior to Anakinra | 15 [15 to 30]
  After Anakinra | 15 [15 to 47]
  At 6 months | 25 [15 to 50]

4. Secondary Outcome: Biologic Efficacy: Inflammation Marker - TNFalpha
Description: Secondary endpoints included the measure of additional inflammatory markers, including TNFalpha.
Time Frame: 6 months post treatment
Population: Patients
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Anakinra Arm
Number analyzed (Participants) | 10
pg/mL
  Prior to Anakinra | 4 [4 to 6]
  After Anakinra | 9 [4 to 30]
  At 6 months | 4 [4 to 33]

ADVERSE EVENTS:
Arm/Group | Anakinra Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No